CLINICAL TRIAL: NCT02577978
Title: Stability of the Medial Pivot Total Knee Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David W. Manning, Associate Professor, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU00090745
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medacta Sphere (Other): Ball-and-socket
  Interventions: Device: Medacta GMK Sphere prosthesis
- Medacta PS (Other): Cam-and-post
  Interventions: Device: Medacta GMK posterior stabilized prosthesis

INTERVENTIONS:
Device: Medacta GMK posterior stabilized prosthesis
  Arms: Medacta PS
Device: Medacta GMK Sphere prosthesis
  Arms: Medacta Sphere

SUMMARY:
The purpose of this study is to compare objective and subjective measures of knee stability following total knee arthroplasty with a medial pivot design vs. a posterior stabilized design.

DETAILED DESCRIPTION:
Several different prostheses are available for use in total knee arthroplasty (TKA). These designs aim to replicate the normal kinematics of the knee joint while maintaining stability throughout a full range of motion. The posterior cruciate ligament (PCL) contributes to these functions in the native knee, and if preserved it can function similarly in the prosthetic knee. Prostheses in which the PCL is sacrificed, and its function not replaced by other means, have poorer outcomes. However, various problems with preserving the PCL, including PCL deterioration in arthritic knees and difficulties with proper tensioning, have led to the development of alternative ways to emulate normal femoral rollback and sagittal plane stability. These posterior-substituted (PS) designs substitute for the PCL with either a cam and post mechanism or a symmetrical ultra-congruent tibial insert.

The cruciate-retaining (CR) and PS designs, together with advances in surgical techniques and component materials, have achieved excellent implant survivorship with rates of > 90% at 20 years. Reports of functional outcomes, however, have been variable. One potential area for improvement in TKA is optimization of implant design to better approximate native knee kinematics. In the normal knee, the medial condyle remains stable in the sagittal plane, functioning like a ball-and-socket, whereas the lateral condyle translates anterior to posterior during flexion. The designs of the CR and PS knees do not allow for this medial-centered rotation. Analysis has revealed paradoxical anterior sliding of the femur during flexion, abnormal axial rotation, and condylar lift-off. Edge loading and increased sagittal plane motion may predispose to accelerated polyethylene wear. The posterior stabilized design uses a cam-and-post mechanism in which one piece of the prosthesis has a plastic post that fits into a slot in the other piece of the prosthesis.

A newer design that attempts to address these issues is the medial pivot knee (MP). This design is characterized by an asymmetrical tibial insert in which the medial compartment is ultra-congruent, providing antero-posterior stability and the lateral compartment allows for rollback around a medial axis of rotation i.e uses a ball-and-socket mechanism. This design more accurately recreates normal knee kinematics, reduces anteroposterior instability, and avoids condylar lift-off. Early studies indicate improved polyethylene wear characteristics. Midterm studies report excellent implant survivorship and clinical outcomes.

Several randomized trials have compared the MP knee favorably with other designs. Patients with bilateral TKAs with a different prosthesis on each side preferred their medial pivot knee to a PS, CR, or mobile-bearing (MB) design. A trial comparing the MP and PS designs found greater range of motion (ROM) and better patient-reported outcomes in the MP group at 2 years. There also exists literature reporting poorer outcomes with the MP design. A trial involving 96 patients who had received both an MP knee and an MB knee on contralateral sides found lower ROM, higher complication rates, and worse patient reported outcomes in the MP knee.

Given the lack of consensus in the literature, further investigation is warranted to determine the impact of the MP design on outcomes following TKA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85, regardless of gender, ethnicity, or pathology
* Must require a total knee arthroplasty
* All subjects must have given signed, informed consent prior to registration in study.

Exclusion Criteria:

* Minors
* Any patients that are unable to consent
* Patients with active infection or osseous tumor of the operative extremity
* Patients undergoing revision surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Department of Orthopaedic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medacta Sphere: Ball-and-socket
  Medacta GMK Sphere prosthesis
- Medacta PS: Cam-and-post
  Medacta GMK posterior stabilized prosthesis
Period: Overall Study
Arm/Group | Medacta Sphere | Medacta PS
Started | 32 | 29
Completed | 25 | 25
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Population: From the total 61 patients enrolled, 11 patients (7 sphere, 4 PS) were dropped from the study due to loss to follow-up. The remainder 50 had data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Medacta Sphere | Medacta PS | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 64 (7) | 66 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (5.82) | 34.2 (5.81) | 33.5 (5.81)
Pre-Operative Ambulatory Status [Count of Participants; unit: Participants] — Patient's ability to ambulate unassisted or assisted with a gait aid
  Participants
    Unassisted | 11 | 16 | 27
    Cane | 10 | 6 | 16
    Walker | 4 | 3 | 7
Hypertension [Count of Participants; unit: Participants] — Patients with a medical history significant for hypertension
  Participants | 20 | 18 | 38
Diabetes Mellitus [Count of Participants; unit: Participants] — Patients with medical history significant for diabetes mellitus
  Participants | 3 | 6 | 9
History of VTE [Count of Participants; unit: Participants] — Patients with medical history significant for venous thromboembolism (VTE)
  Participants | 4 | 1 | 5
Pre-operative Narcotic Use [Count of Participants; unit: Participants] — Patients with recent history of narcotic use for pain management prior to surgery
  Participants | 4 | 4 | 8
Tobacco Use [Count of Participants; unit: Participants] — Patients with active or recent tobacco use prior to surgery
  Participants | 3 | 5 | 8
Coronary Artery Disease [Count of Participants; unit: Participants] — Patients with medical history significant for coronary artery disease
  Participants | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score (OKS) Pre-operative Through 2 Years Post-operative
Description: Patient completed Oxford Knee Score questionnaire used to assess the patient's perspective of outcome following Total Knee Arthroplasty (TKA); score range is reported between 0-48 with improvement in outcomes reflected as a higher numerical value (e.g. a 'complete' return to pre-disease functionality would be reported as a score of 48)
Time Frame: Pre-operatively on day of surgery, 6 weeks, 3 months, 6 months, 12 months and 24 months post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline Oxford Knee Score | 16.31 (7.66) | 19.88 (9.39)
  6 wk. Post Op Oxford Knee Score | 29.96 (9.64) | 28.52 (8.77)
  3 mo. Post Op Oxford Knee Score | 32.0 (11.35) | 32.7 (9.47)
  6 mo. Post Op Oxford Knee Score | 33.67 (8.9) | 36.41 (10.58)
  1 yr. Post Op Oxford Knee Score | 39.16 (9.97) | 35.81 (11.33)
  2 yr. Post Op Oxford Knee Score | 40.41 (8.56) | 38.28 (11.8)

2. Primary Outcome: Veteran's RAND 12 (VR-12) Mental Composite Score (MCS) Through 2 Years Post Operative
Description: Veteran's RAND 12 Item Health Survey used to assess health-related quality of life, to estimate disease burden, and to evaluate disease-specific benchmarks. Scores for the Mental Composite Score (MCS) range from 5.2 to 76.3 and are evaluated as a summative T-score with population mean of 50 (Standard Deviation = 10);higher scores indicate improved mental wellness/function as reported by patients.
Time Frame: Pre-operatively, 6 weeks post-operatively, 3 months post-operatively, 6 months post-operatively, 12 months post-operatively, and 2 years post-operatively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline VR-12 MCS | 44.97 (14.13) | 54.33 (12.35)
  6 wk. VR-12 MCS | 49.25 (14.69) | 59 (7.18)
  3 mo. VR-12 MCS | 51.11 (11.74) | 53.71 (12.71)
  6 mo. VR-12 MCS | 53.6 (11.79) | 53.85 (10.75)
  1 yr. VR-12 MCS | 53.7 (11.22) | 54.09 (12.47)
  2 yr. VR-12 MCS | 54.83 (9.54) | 54.78 (10.27)

3. Primary Outcome: Veteran's RAND 12 (VR-12) Physical Composite Score (PCS) Through 2 Years Post Operative
Description: Veteran's RAND 12 Item Health Survey used to assess health-related quality of life, to estimate disease burden, and to evaluate disease-specific benchmarks. Scores for the Physical Composite Score (MCS) range from 6.3 to 71.8 and are evaluated as a summative T-score with population mean of 50 (Standard Deviation = 10);higher scores indicate improved physical wellness/function as reported by patients.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline VR-12 PCS | 26.74 (8.3) | 23.92 (6.71)
  6 wk. VR-12 PCS | 34.5 (8.1) | 34.02 (11.1)
  3 mo. VR-12 PCS | 38.27 (12.58) | 35.9 (10.28)
  6 mo. VR-12 PCS | 39.5 (10.23) | 42.1 (11.25)
  1 yr. VR-12 PCS | 46.36 (12.22) | 42.48 (12.54)
  2 yr. VR-12 PCS | 42.76 (11.08) | 46.01 (12.85)

4. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Physical Function Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Physical Function domain higher scores indicated improved physical function as reported by the patient
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline PROMIS Physical Function | 32.92 (4.44) | 31.24 (5.27)
  6 wk. PROMIS Physical Function | 38.38 (6.95) | 39.96 (6.45)
  3 mo. PROMIS Physical Function | 42.12 (8.14) | 41.32 (6.76)
  6 mo. PROMIS Physical Function | 43.81 (7.26) | 45.36 (9.09)
  1 yr. PROMIS Physical Function | 48.06 (9.22) | 48.9 (10.25)
  2 yr. PROMIS Physical Function | 49.17 (7.84) | 46.5 (8.97)

5. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Pain Interference Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Pain Interference domain an increased value indicates greater severity/frequency of pain reported by the patient.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline PROMIS Pain Interference | 66.03 (4.73) | 65.88 (7.39)
  6 wk. PROMIS Pain Interference | 58.23 (8.59) | 58.2 (7.62)
  3 mo. PROMIS Pain Interference | 55.9 (11.48) | 55.53 (9.9)
  6 mo. PROMIS Pain Interference | 52.83 (9.31) | 53.27 (12.35)
  1 yr. PROMIS Pain Interference | 46.65 (11.22) | 49.98 (11.22)
  2 yr. PROMIS Pain Interference | 44.7 (8.63) | 46.97 (10.96)

6. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Pain Behavior Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Pain Behavior domain an increased value indicates greater severity/frequency of pain reported by the patient
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline PROMIS Pain Behavior | 60.98 (3.22) | 60.92 (4.88)
  6 wk. PROMIS Pain Behavior | 56.79 (7.27) | 58.49 (3.6)
  3 mo. PROMIS Pain Behavior | 54.14 (7.78) | 53.6 (9.41)
  6 mo. PROMIS Pain Behavior | 53.2 (8.72) | 51.25 (9.27)
  1 yr. PROMIS Pain Behavior | 45.92 (11.31) | 47.95 (12.43)
  2 yr. PROMIS Pain Behavior | 42.76 (9.09) | 46.29 (10.36)

7. Primary Outcome: Total Score Calculated Using the Forgotten Joint Score in Order to Assess the Subject's Ability to Forget the Artificial Joint in Everyday Life
Description: Patient completed questionnaire used to assess the patients' ability to forget about a joint as a result of successful treatment. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60 where a high score indicates an improved outcome. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score with higher scores indicating improved physical function/reduced impact of symptoms on activity:
  Final score = 100 - ((sum(item01 to item12) - 12)/48*100)
Time Frame: 12 months post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale | 57.1 (37.6) | 54.6 (41.6)

8. Primary Outcome: International Knee Documentation Committee (IKDC) Questionnaire Assessed Through 2 Years Post-op
Description: The International Knee Documentation Committe (IKDC) Questionnaire is a subjective scale that provides patients with an overall function score based on a summative score for 3 sub categories (knee function, sports activities, pain/symptoms). A score between 0-100 is obtained as the sum of scores for each individual question, with increasing composite scores correlating positively with patient functional status/quality of life.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline IKDC Composite | 35.82 (8.72) | 35.97 (6.97)
  6 wk. IKDC Composite | 42.38 (11.19) | 43.91 (7.68)
  3 mo. IKDC Composite | 50.41 (11.44) | 44.5 (10.4)
  6 mo. IKDC Composite | 48.72 (12.08) | 48.52 (11.73)
  1 yr. IKDC Composite | 57.97 (13.79) | 52.66 (13.23)
  2 yr. IKDC Composite | 51.26 (8.67) | 49.3 (10.56)

9. Primary Outcome: Score for the Knee Society Score (KSS) Knee Component at 1 Year Post-operatively
Description: Physician completed Knee Society Score questionnaire used to measure a patient's functional ability before and after total knee arthroplasty (TKA); score range is reported between 0-100 with improvement in outcomes reflected as a higher numerical value (e.g. a 'complete' return to pre-disease functionality would be reported as a score of 100)
Time Frame: 12 months post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale | 88.1 (9.5) | 86.0 (12.6)

10. Primary Outcome: Score for the Knee Society Score (KSS) Function Component at 1 Year Post-operatively
Description: as for outcome 9
Time Frame: 12 months post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
score on a scale | 81.4 (17.9) | 77.4 (22.5)

11. Secondary Outcome: Assessing Knee Stability Using the KT-1000 Arthrometer (at 30 Degrees)
Description: Used for grading the stability of the knee in various degrees of flexion according to section 4 of the International Knee Documentation Committee's Knee Ligament Standard Evaluation Form where normal (-1 to 2 mm); nearly normal (3 to 5 mm); abnormal (6 to 10 mm); severely abnormal (>10 mm)
Time Frame: 1 year post-operatively
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
millimeters | 5.6 (1.9) | 10.2 (2.7)

12. Secondary Outcome: Assessing Knee Stability Using the KT-1000 Arthrometer (at 90 Degrees)
Description: as for outcome 11
Time Frame: 1 year post-operatively
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
millimeters | 4.1 (2.0) | 5.6 (1.9)

13. Secondary Outcome: Get-up-and-Go Test
Description: Used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down.
Time Frame: Between 6 months and 1 year post-operatively
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Medacta Sphere | Medacta PS
Number analyzed (Participants) | 25 | 25
seconds | 10.2 (3.7) | 10.5 (5.0)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Medacta Sphere | Medacta PS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02577978/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02577978/ICF_001.pdf